CLINICAL TRIAL: NCT03249285
Title: Pharmacogenomics Of Hypertension: A New Approach For A Personalized Medicine
Brief Title: Pharmacogenomics of Hypertension Personalized Medicine (PGX-HT)
Acronym: PGX-HT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Chiara Lanzani, medical doctor, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: udraCT NUMBER: 2015-001888-39
Record Dates: First submitted 2017-02-13; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Hypertension
Keywords: hypertension; pharmacogenomics; anti-hypertensive therapy
MeSH Terms: conditions — Hypertension | interventions — Perindopril; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Peri profile yes (Experimental): patient with genetic Perindopril profile, receiving Perindopril treatment with 4-8 mg/day oral for 4-8 weeks
  Interventions: Drug: Peri
- HCTZ profile yes (Experimental): patient with genetic HCTZ profile, receiving HCTZ treatment with 12,5-25 mg/day oral for 4-8 weeks
  Interventions: Drug: HCTZ
- Peri no profile (Active Comparator): patient with no genetic profile, receiving after randomisation Perindopril treatment with 4-8 mg/day oral for 4-8 weeks
  Interventions: Drug: Peri
- HCTZ no profile (Active Comparator): patient with no genetic profile, receiving after randomisation HCTZ treatment with 12,5-25 mg/day oral for 4-8 weeks
  Interventions: Drug: HCTZ

INTERVENTIONS:
Drug: Peri — Perindopril 4 mg /day, orally with titration to 8 mg/day after 1 month if BP (Blood pressure) is not controlled
  Other Names: Perindopril
  Arms: Peri no profile; Peri profile yes
Drug: HCTZ — Hydrochlorothiazide 12, 5 mg day, orally with titration to 25 mg/day after 1 month if BP is not controlled
  Other Names: Hydrochlorothiazide
  Arms: HCTZ no profile; HCTZ profile yes

SUMMARY:
This is a pharmacogenomic prospective , four-arms, parallel groups, active comparator controlled study in essential hypertensive patients never treated before.

Each patient will be genotyped for SNPs (single nucleotide polymorphism) in preliminary genetic profiles and will be treated according to their genetic profile with Peri (Perindopril) 4 mg or HCTZ ( hydrochlorothiazide) 12.5 mg.

DETAILED DESCRIPTION:
At screening visit each patient will be genotyped for SNPs in preliminary genetic profiles with a custom SNP array.

The therapy scheme includes 2-4-week run-in period after which eligible patients will be treated according to their genetic profile with Peri 4 mg or HCTZ 12.5 mg. Titration to Peri 8 mg or HCTZ 25 mg could be possible after one month treatment.

Patients without any genetic profile will be randomly assigned to HCTZ or Peri treatment as control groups.

The treatment period will last 8 weeks, while the study about 10-12 weeks

Four cases may occur:

* patient with HCTZ profile, HCTZ treatment;
* patient with Peri profile, Peri treatment;
* patient without HCTZ nor Peri profile, randomization for HCTZ or Peri;
* patient with both profiles, treatment according to the profile with the higher number of positive contributors.

Eligible patients will be treated according to their genetic profile with Peri 4 mg or HCTZ 12.5 mg/die.

Titration to Peri 8 mg or HCTZ 25 mg could be possible after 4 weeks treatment. The treatment period will last 8 weeks, while the study about 10-12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male/Female patients aged 25-60 years.
* Naive hypertensive patients (newly diagnosed, never treated before).
* Documented mild to moderate arterial hypertension, as defined below:

  1. At Visits 1 and 2 (week -4 and week -2 run-in period) the mean of the last 3 consecutive readings of office SBP must be >= 140 mmHg and/or DBP must be >=90 mmHg, when measured by office blood pressure (OBP);
  2. At Visit 3 (week 0) enrolment , the mean of the last 3 consecutive readings of SBP must be >= 140 mmHg and <160 mmHg, and DBP must be >= 90 mmHg and <110 mmHg, when measured by OBP.
* Signed informed consent for genotyping.

Exclusion Criteria:

* known causes of secondary hypertension;
* pregnant, nursing women or women of childbearing potential taking anti-contraceptive medication;
* severe or malignant hypertension;
* history of renal artery disease;
* significant renal disease (estimated creatinine clearance less than 60 mL/min);
* hepatic disease;
* cardiac diseases (myocardial infarction, atrial fibrillation, etc);
* diabetes (fasting plasma glucose >125mg/dL);
* statin treatment;
* obesity (BMI>30 kg/m2).

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
SBP (Systolic blood pressure) and DBP (Diastolic blood pressure) response | 4 and 8 weeks
  Difference in SBP and DBP variation after 4 and 8 weeks of therapy according to the presence or not of specific genetic profile for each drugs

SECONDARY OUTCOMES:
Profiles implementation | in the three months after the end of the study
  Implementing and redefining the genetic profile for HCTZ or/and Peri by using a further spectrum of 128 different SNP variants

CONTACTS AND LOCATIONS:
Overall Officials: Manunta Paolo, Professor, Study Chair — Scientif Institute San Raffale
Locations (3):
- Italy (3):
  - Azienda Sanitaria 6, Livorno
  - San Raffaele Hospital, Milan
  - Azienda Ospedaliero - Universitaria S. Maria della Misericordia, Udine

IPD SHARING:
Plan to Share IPD: Undecided